CLINICAL TRIAL: NCT00142259
Title: Randomisierte, Doppelblinde Langzeitstudie Zur Klinischen Wirksamkeit Der Bilateralen Globus Pallidus Internus-Stimulation Bei Idiopathischer Generalisierter Oder Segmentaler Dystonie
Brief Title: Efficacy and Safety of DBS of the GPi in Patients With Primary Generalized and Segmental Dystonia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: German Parkinson Study Group (GPS) (Other)
Collaborators: Medtronic (Industry); Competence Network on Parkinson's Disease (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15; Grant: 01 GI 0201 / 01 GI 0401
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2006-12-06 (Estimated); Status verified 2005-09

CONDITIONS: Dystonia
Keywords: deep brain stimulation; internal globus pallidus; dystonia
MeSH Terms: conditions — Dystonia

INTERVENTIONS:
Device: Deep brain stimulation of the internal globus pallidus

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of bilateral deep brain stimulation of the internal globus pallidus for treating idiopathic generalized or severe segmental dystonia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic multifocal, segmental or generalised dystonia
* duration of disease > 5 years
* age between 14 and 75 years
* relevant disability in activities of daily living despite optimal drug treatment
* informed consent signed by the patient
* For adolescents between 14 and 18 years: an additional informed consent signed by a legal guardian is necessary

Exclusion Criteria:

* Mattis-Score < 120
* BDI > 25
* previous stereotactic brain surgery
* severe brain atrophy
* increased bleeding risk
* immunosuppression and increased risk of infection
* relevant cerebrovascular disease
* psychiatric disorders, which might interfere with the cooperation in the study
* other contraindications for surgery

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2002-10; Study Completion 2009-08

PRIMARY OUTCOMES:
relative change of the individual Burk-Fahn-Marsden-Dystonia motor score 3 months after treatment compared to baseline

SECONDARY OUTCOMES:
relative change of the individual Burk-Fahn-Marsden-Dystonia ADL score 3 months after treatment compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jens Volkmann, MD, PhD, Principal Investigator — Dept. Neurology, UKSH Campus Kiel, Germany
Locations (8):
- Medical University Innsbruck, Department of Neurology, Innsbruck, Tyrol, Austria
- Germany (7):
  - Klinikum der LMU, Neurologische Klinik, München, Bavaria
  - Neurologische Klinik am Klinikum der BJM-Universität, Würzburg, Bavaria
  - Department of Neurology, Charité, Humboldt-University Berlin, Berlin, State of Berlin
  - Düsseldorf
  - Department of Neurology, University Heidelberg, Heidelberg
  - Dept. Neurology, UKSH Campus Kiel, Kiel
  - Department of Neurology, University Rostock, Rostock

REFERENCES:
- [Result] Kupsch A, Benecke R, Muller J, Trottenberg T, Schneider GH, Poewe W, Eisner W, Wolters A, Muller JU, Deuschl G, Pinsker MO, Skogseid IM, Roeste GK, Vollmer-Haase J, Brentrup A, Krause M, Tronnier V, Schnitzler A, Voges J, Nikkhah G, Vesper J, Naumann M, Volkmann J; Deep-Brain Stimulation for Dystonia Study Group. Pallidal deep-brain stimulation in primary generalized or segmental dystonia. N Engl J Med. 2006 Nov 9;355(19):1978-90. doi: 10.1056/NEJMoa063618. PMID 17093249
- [Derived] Steigerwald F, Kirsch AD, Kuhn AA, Kupsch A, Mueller J, Eisner W, Deuschl G, Falk D, Schnitzler A, Skogseid IM, Vollmer-Haase J, Ip CW, Tronnier V, Vesper J, Naumann M, Volkmann J; DBS study group for dystonia. Evaluation of a programming algorithm for deep brain stimulation in dystonia used in a double-blind, sham-controlled multicenter study. Neurol Res Pract. 2019 Sep 24;1:25. doi: 10.1186/s42466-019-0032-2. eCollection 2019. PMID 33324891
- [Derived] Volkmann J, Wolters A, Kupsch A, Muller J, Kuhn AA, Schneider GH, Poewe W, Hering S, Eisner W, Muller JU, Deuschl G, Pinsker MO, Skogseid IM, Roeste GK, Krause M, Tronnier V, Schnitzler A, Voges J, Nikkhah G, Vesper J, Classen J, Naumann M, Benecke R; DBS study group for dystonia. Pallidal deep brain stimulation in patients with primary generalised or segmental dystonia: 5-year follow-up of a randomised trial. Lancet Neurol. 2012 Dec;11(12):1029-38. doi: 10.1016/S1474-4422(12)70257-0. Epub 2012 Nov 1. PMID 23123071
- See also: Homepage Competence Network on Parkinson's disease sponsored by the German government — http://www.kompetenznetz-parkinson.de